CLINICAL TRIAL: NCT04188132
Title: EEG Based Brain Computer Interface in Chronic Stroke Survivors for Upper Limb Rehabilitation- A Pilot Study Using Motor Execution and Motor Imagery
Brief Title: EEG Based BCI for Upper Limb Rehabilitation in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Subasree Ramakrishnan, Visiting Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001846
Record Dates: First submitted 2019-10-28; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Stroke Sequelae; Brain Ischemia
MeSH Terms: conditions — Brain Ischemia | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Pilot study in patients with fulfilling the eligibility criteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG BCI closed loop feedback for rehabilitation of upper limb (Experimental): This study is a pilot study to examine the feasibility of a SMR based EEG BCI using motor task and motor imagery and involve a gaming feedback for same.
  The first two days will be used for calibrating the BMI using commands in computer screen followed by further two days for testing the BMI and feedback control during gaming in computer to move the ball in the computer screen.
  Interventions: Other: EEG -BCI based Feedback for rehabilitation

INTERVENTIONS:
Other: EEG -BCI based Feedback for rehabilitation — Subjects will undergo EEG based BCI as feedback for rehabilitation

SUMMARY:
Biomedical and Engineering approaches form a key element to neurological rehabilitation of upper limbs. Brain Computer Interface (BCI) using Motor execution and Motor Imagery are known to aid motor recovery in stroke. The purpose of this study is to demonstrate that Noninvasive Sensorimotor Rhythm (SMR) based EEG based BCI using motor execution and Motor Imagery tasks can aid in rehabilitation of upper limb movements in chronic stroke.

The project aims to explore an SMR-based BCI system that can exploit the sensorimotor rhythm voluntary modulation to play a virtual game as neurofeedback using motor executory tasks and imagined hand movements by stroke patients, who suffer from upper limb disability.

DETAILED DESCRIPTION:
Brain Computer Interface (BCI) using Motor execution and Motor Imagery are known to aid motor recovery in stroke. The purpose of this study is to demonstrate that Noninvasive Sensorimotor Rhythm (SMR) based EEG based BCI using motor execution and Motor Imagery tasks can aid in rehabilitation of upper limb movements in chronic stroke.

The project aims to explore an SMR-based BCI system that can exploit the sensorimotor rhythm voluntary modulation to play a virtual game as neurofeedback using motor executory tasks and imagined hand movements by stroke patients, who suffer from upper limb disability. Studies have shown that movement and motor imagery (MI) (i.e., the mental rehearsal of a movement without any activation of the muscles) induce similar EEG patterns over the motor cortex.

Movement execution, preparation and even observation are usually accompanied by a decrease in µ- and β-rhythm in the cortical area representing the involved body segment. Such a reduction is called event-related desynchronization (ERD).The increase in µ-rhythm, i.e. event-related synchronization (ERS), is observed in the regions of the brain representing body segments, which are not involved in the task.This study is a pilot study to examine the feasibility of a SMR based EEG BCI using motor task and motor imagery and involve a gaming feedback for same.

The first two days will be used for calibrating the BMI using commands in computer screen followed by further two days for testing the BMI and feedback control during gaming in computer to move the ball in the computer screen.

ELIGIBILITY:
Inclusion Criteria:

* • age: 21-75 years

  * Subacute or chronic stroke; interval of at least 3 months and interval of at least 6 months from stroke to time of enrollment, respectively.
  * no cerebellar signs or bilateral motor deficit
  * Cognitive ability to consent, assimilate, and participate actively in the treatment protocol (Mini Mental State Examination score > 24 points, out of a total 30 indicating normal cognitive ability);
  * Modified Rankin scale scores 1-3 (Mild-Moderate functional disability post-stroke);
  * Modified Ashworth Scale of Spasticity score <= 3 (ranges from 0-4 with 4 reflecting maximum spasticity)
  * No epilepsy /usage of antiepileptic drug

    ◦ Subjects with Stroke will be included if they have:
  * unilateral impaired upper limb
  * Able to initiate hand movements like opening and closing fist and no joint contracture or severe spasticity in the affected upper limbs.
  * Sufficient sitting balance to participate in experimental activities.
  * No condition (e.g. severe arthritis, central pain) that would interfere with the administration of motor function tests.
  * English-language comprehension and cognitive ability sufficient to give informed consent (MMSE >=24) and to cooperate with the intervention.

Exclusion Criteria:

* • Orthopedic conditions of either upper or lower extremity that would affect performance on the study

  * untreated depression that may affect motivation to participate in the study
  * vascular cognitive impairment interfering with comprehending the tasks
  * Individuals with stroke who have been diagnosed with cognitive or severe visual deficits, hemineglect, uncontrolled angina, or pregnancy
  * no psychiatric or neurological condition other than stroke

    ◦ Stroke will be excluded if they have:
  * Pregnancy (Self -reported)
  * Dementia (MMSE score less than 24)
  * Recurrence of stroke (Occurrence of new focal deficits reported by patient or detected by PI on examination during visits)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment score (Upper limb)(Min0-Max66;Total 66) | 4 days
  Change in Hand strength
Decoding motor intent of hand movements using Scalp Electroencephalography(EEG) | 4 days
  Electroencephalographic spectral power changes during Motor execution and Motor Imagery of hand movements in stroke subjects

CONTACTS AND LOCATIONS:
Overall Officials: Subasree R, Principal Investigator — University of Houston
Locations (1):
- Subasree Ramakrishnan, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Currently not planning for data sharing

REFERENCES:
- [Background] Daly JJ, Wolpaw JR. Brain-computer interfaces in neurological rehabilitation. Lancet Neurol. 2008 Nov;7(11):1032-43. doi: 10.1016/S1474-4422(08)70223-0. Epub 2008 Oct 2. PMID 18835541
- [Background] Ramos-Murguialday A, Broetz D, Rea M, Laer L, Yilmaz O, Brasil FL, Liberati G, Curado MR, Garcia-Cossio E, Vyziotis A, Cho W, Agostini M, Soares E, Soekadar S, Caria A, Cohen LG, Birbaumer N. Brain-machine interface in chronic stroke rehabilitation: a controlled study. Ann Neurol. 2013 Jul;74(1):100-8. doi: 10.1002/ana.23879. Epub 2013 Aug 7. PMID 23494615